CLINICAL TRIAL: NCT01869374
Title: Improving Outcomes in Geriatric Depression: Magnetic Seizure Therapy
Brief Title: Study Comparing Magnetic Seizure Therapy (MST) to Electroconvulsive Therapy (ECT) for Depression in Older Adults
Acronym: MSTvsEST
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Stefan Rowny, Assistant Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6427
Record Dates: First submitted 2013-05-22; First posted 2013-06-05 (Estimated); Results first posted 2020-06-19 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-08

CONDITIONS: Depression; Major Depressive Episode; Bipolar Disorder
Keywords: Depression; Brain Stimulation; Seizure therapy; Convulsive Therapy
MeSH Terms: conditions — Depression; Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: Electroconvulsive Therapy / Magnetic Seizure Therapy
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnetic Seizure Therapy (MST) (Experimental): MagVenture MagPro MST device
  Interventions: Device: MagVenture MagPro MST
- RUL ECT (Active Comparator): Right Unilateral ECT with the Somatics Thymatron device using Ultrabrief stimulus
  Interventions: Biological: RUL ECT

INTERVENTIONS:
Device: MagVenture MagPro MST — Brain stimulation by magnetic means versus electrical standard unilateral Electroconvulsive Therapy (RUL ECT). Treatment will be administered 3 times a week.
  Arms: Magnetic Seizure Therapy (MST)
Biological: RUL ECT — RUL ECT using the Somatics Thymatron device with Ultrabrief stimulus. Treatment will be administered 3 times a week.
  Other Names: Right Unilateral Electroconvulsive Therapy
  Arms: RUL ECT

SUMMARY:
To evaluate the feasibility, tolerability and efficacy of Magnetic Seizure Therapy (MST) in elderly patients with a major depressive episode, who are randomly assigned to receive an acute course of MST or ECT.

The investigators hypothesize:

1. MST and ECT will have similar antidepressant efficacy
2. MST will have less post-treatment amnesia than ECT as reflected in a primary measures of anterograde and retrograde amnesia following the acute treatment phase.
3. At follow up, MST will show a lesser degree of persisting deficit in measures of retrograde amnesia than ECT.

DETAILED DESCRIPTION:
The purpose of this study is to compare the clinical efficacy and side effects of Magnetic Seizure Therapy (MST) and Electroconvulsive Therapy (ECT) in older adults currently experiencing a major depressive episode in the context of either unipolar or bipolar depression. ECT is known to be highly effective in treating depression, but it can have some adverse cognitive side effects. MST is a new form of convulsive therapy that is being developed as a means of improving the side effect profile of ECT so that more patients may benefit without suffering significant detrimental effects on cognition.

Both ECT and MST rely on a therapeutic seizure, but they do so in different ways. In ECT, an electrical stimulator is used to pass electrical current between two electrodes placed on the surface of person's head, which causes some electricity to go through the brain and cause a seizure. In MST, a magnetic stimulator is used to create a magnetic field in a targeted area of the brain, which induces a small electrical field in the neurons that causes a seizure. Treatments will be administered three times a week.

In addition to the treatment sessions, this study will involve a number of assessments at different time-points (i.e., baseline prior to treatment, post-treatment, 2 months post-treatment and 6 months post-treatment) that are used to evaluate the person's antidepressant response and the physical and cognitive side effects of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 55-90
* Clinical diagnosis of major depressive episode, in the context of unipolar or bipolar disorder
* Willing and capable to provide informed consent
* Convulsive therapy clinically indicated
* Hamilton Rating Scale for Depression (HRSD24)≥ 20
* Mini Mental State Exam (MMSE) ≥ 24
* For outpatients: responsible adult living with the patient

Exclusion Criteria:

* Current unstable or serious medical condition, or any comorbid medical condition that substantially increases the risks of ECT (such as acute myocardial infarction, space occupying brain lesion or other cause of increased intracranial pressure, unstable aneurysm or vascular malformation, poorly controlled diabetes mellitus, carcinoma, renal failure, hepatic failure)
* History of neurological disorder, epilepsy, stroke, brain surgery, metal in the head, history of known structural brain lesion
* Presence of devices that may be affected by MST (pacemaker, medication pump, cochlear implant, implanted brain stimulator, or vagus nerve stimulator implanted)
* History of head trauma with loss of consciousness for greater than 5 minutes
* History of schizophrenia, schizoaffective disorder, or rapid cycling bipolar disorder
* History of substance abuse or dependence in past 3 months
* Failure to respond to an adequate course of ECT in the current depressive episode
* History of ECT in the past 6 months and/or failure to respond to an adequate trial of ECT lifetime
* Presence of intracardiac lines

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2020-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan B Rowny, MD, MFA, Principal Investigator — NYSPI/Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rowny, S., & Lisanby, S. H. (2009). Other Brain Stimulation Methods. In B. J. Sadock, V.A. Sadock & P. Ruiz (Eds.) . Kaplan and Sadock's Comprehensive Textbook of Psychiatry (9th ed.) (Pp. 3301-3314). Lippincott Williams & Wilkins. Philadelphia:PA.
- [Background] Rowny SB, Benzl K, Lisanby SH. Translational development strategy for magnetic seizure therapy. Exp Neurol. 2009 Sep;219(1):27-35. doi: 10.1016/j.expneurol.2009.03.029. Epub 2009 Apr 5. PMID 19348798
- [Background] McClintock SM, DeWind NK, Husain MM, Rowny SB, Spellman TJ, Terrace H, Lisanby SH. Disruption of component processes of spatial working memory by electroconvulsive shock but not magnetic seizure therapy. Int J Neuropsychopharmacol. 2013 Feb;16(1):177-87. doi: 10.1017/S1461145711001866. Epub 2012 Jan 5. PMID 22217479
- [Background] Rowny SB, Cycowicz YM, McClintock SM, Truesdale MD, Luber B, Lisanby SH. Differential heart rate response to magnetic seizure therapy (MST) relative to electroconvulsive therapy: a nonhuman primate model. Neuroimage. 2009 Sep;47(3):1086-91. doi: 10.1016/j.neuroimage.2009.05.070. Epub 2009 Jun 2. PMID 19497373
- [Background] Rowny, S., & Lisanby, S. H. (2008). Brain Stimulation in Psychiatry. In A. Tasman, J. Kay, J. A. Lieberman, M. B. First & M. Maj (Eds.), Psychiatry (3rd ed.) (pp.2354-2371). Chichester, UK: John Wiley & Sons. DOI: 10.1002/9780470515167.ch109
- [Derived] Jiang J, Zhang C, Li C, Chen Z, Cao X, Wang H, Li W, Wang J. Magnetic seizure therapy for treatment-resistant depression. Cochrane Database Syst Rev. 2021 Jun 16;6(6):CD013528. doi: 10.1002/14651858.CD013528.pub2. PMID 34131914

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Five-day washout from all anti-depressants and mood stabilizers.
Period: Overall Study
Arm/Group | Magnetic Seizure Therapy (MST) | RUL ECT
Started | 9 | 9
Completed | 9 | 8
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Right Unilateral ECT (RUL ECT): Right Unilateral ECT with the Somatics Thymatron device using Ultrabrief stimulus
  RUL ECT: RUL ECT using the Somatics Thymatron device with Ultrabrief stimulus. Treatment will be administered 3 times a week.
- Total: Total of all reporting groups
Arm/Group | Magnetic Seizure Therapy (MST) | Right Unilateral ECT (RUL ECT) | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 4 | 9
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Full Range); unit: years] | 66.3 [56 to 79] | 65.3 [58 to 74] | 65.8 [56 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 3 | 4 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression, 24-Item (HRSD-24)
Description: The unabbreviated scale title is "Hamilton Rating Scale for Depression." As its title suggests, this is a clinical measure of major depressive disorder.
  The minimum score a participant could receive on this measure is 0. The maximum score that a participant could receive is 75. Please see a table written below that associates HRSD-24 values with clinical outcome:
  0-7 = no depression 8-16 = mild depression 17-23 = moderate depression 24 and up = severe depression
  Calculation details: Outcome data corresponds to baseline HRSD-24 score subtracted from post-tx HRSD-24 score. The larger difference, therefore, corresponds to the more effective treatment for this study.
Time Frame: baseline (pre-treatment) and post-treatment
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Magnetic Seizure Therapy (MST) | RUL ECT
Number analyzed (Participants) | 9 | 9
units on a scale | 22.625 [16 to 29] | 15.375 [2 to 25]

ADVERSE EVENTS:
Time Frame: Adverse event data for participants was collected from baseline to post-treatment (between two and three months, depending on the participants' number of treatments).
Description: This study did not include a design for monitoring or assessing adverse events. We did not consider any of our participants to be at risk of serious adverse events or all-cause mortality. Prior to enrollment in the study, all our participants were evaluated by a physician and anesthesiologist and were medically cleared to receive an acute course of convulsive therapy. Any risk that would have been contraindicated with convulsive therapy was ruled out in advance of participants' pre-tx scan.
Arm/Group | Magnetic Seizure Therapy (MST) | RUL ECT
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2016-07-28): https://cdn.clinicaltrials.gov/large-docs/74/NCT01869374/ICF_000.pdf
  • Study Protocol (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT01869374/Prot_001.pdf